CLINICAL TRIAL: NCT05970146
Title: Comparison Between Cervical Epidural and Stellate Ganglion Block in Management of Complex Regional Pain Syndrome of the Upper Limb A Prospective Comparative Study
Brief Title: Cervical Epidural and Stellate Ganglion Block in Upper Limb Complex Regional Pain Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Hassan Moustafa Hegazy, Assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264MD58/3/23
Record Dates: First submitted 2023-07-19; First posted 2023-08-01 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Stellate Ganglion Block; Cervical Epidural; Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided Stellate ganglion block (Experimental): The procedure is going to be the anterior paratracheal approach on the cervical sympathetic chain
  Interventions: Drug: Ultrasound guided Stellate ganglion block
- unilateral cervical epidural (Experimental): The patient is placed in prone position, with stabilization of the forehead on a padded support
  Interventions: Drug: unilateral cervical epidural

INTERVENTIONS:
Drug: Ultrasound guided Stellate ganglion block — Under visualization with ultrasound, a 22-gauge, 5-cm needle inserted perpendicular to the skin to rest anteriorly to the precervical fascia. 6 mL lidocaine 0.125% and 8 mg dexamethasone in a total volume of 8 mL is used. After injection of a 0.5-mL test dose to exclude intravascular positioning, the remainder of the appropriate dose was administered. The patient will be encouraged to lie flat for 3 minutes after the injection and then to sit up.
  Arms: Ultrasound guided Stellate ganglion block
Drug: unilateral cervical epidural — Aseptic betadine skin preparation will be performed and sterile drapes will be applied. Local anesthetic infiltration of the skin at C7-T1 interspace will be done using 2-3 mL of lidocaine 2% with guidance of the C-arm an 18-gauge. Tuohy needle will be inserted at C7-T1 interspace and directed towards either right or left epidural recess according to the site of the operation. Identification of entering the epidural space will be confirmed by hanging drop technique. The position of the needle is the confirmed by injection of 1 mL of non-ionized diluted dye (omnipause 300) to confirm unilateral spread of the dye. After that, a test dose was administrated, consisting of 2 mL of 2% lidocaine with 1:200,000 epinephrine.
  Arms: unilateral cervical epidural

SUMMARY:
Evaluate the efficacy of two regimens of management in relieving chronic refractory pain in patients with upper limb complex regional pain syndrome after orthopedic trauma

DETAILED DESCRIPTION:
Ideal therapy for Complex Regional Pain Syndrome is multimodal with the use of physical therapy, psychotherapy, and pharmacologic therapy to complement interventional procedures. Within pharmacotherapy, drugs most often utilized include non steroidal anti-inflammatory drugs (NSAIDs), gamma-aminobutyric acid receptor agonists (i.e., gabapentin, pregabalin), and N-methyl-D-aspartate (NMDA) receptor antagonists (i.e., Ketamine).

In complex Regional Pain Syndrome treatment, stellate ganglion block (SGB) is a well-established method of nerve blockade of the sympathetic ganglia in the lower cervical and upper thoracic region.

Epidural block have differential block as sensory, motor, and sympathetic. Nerve functions are blunt at different rates and to different degrees. Sensory block occurs with a lower concentration of Local anathesia and develops faster than motor block with coexisting sympathectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged more than 21 years old of both sexes with American Society of Anesthesiologists I and II
2. Upper limb trauma patients with pain disproportionate to the degree of tissue injury and persists beyond the normal expected time for tissue healing
3. Patients diagnosed as (Complex Regional Pain Syndrome ) based on Budapest criteria There should be at least one symptom or sign in three of the four previous categories that can not be explained by other diagnosis.
4. The average daily pain intensity required on Numerical Rating Scale is 7 or more for at least 3 months despite of standard therapy which includes: (pharmacologic therapy Non-steroidal anti-inflammatory drugs, Antiepileptic drugs(AEDs), antidepressants), as well as physical therapy and psychiatric care.

Exclusion Criteria:

* Patient refusal
* Patients with unstable psychological or psychiatric conditions, including: untreated bipolar disorder, post-traumatic stress disorder, major depression, severe personality disorder and psychotic illness
* Patients have recently undergone major interventional pain procedures, such as nerve blocks or implantable therapies.
* Patients with known drug dependency or substance use disorder specifically related to ketamine or other psycho-stimulant drugs
* Patients with previous severe reactions, contraindication or allergy to ketamine
* Patients with hepatic or renal impairment
* Active infection at the injection site
* Known allergies to medications
* Previous neck surgeries
* Raynaud's disease or Raynaud's phenomena
* Coagulopathy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The percent on satisfactory relief of pain | 6 month post injection
  Numerical rating scales (NRS) is an 11-Point Scale for patient self-reporting of pain. It is based solely on the ability to perform activities of daily living (ADLs) with 0 being "no pain" and 10 being "the worst pain imaginable.
  NRS was measured before, immediately after injection, 3 and 6 month post injection.

SECONDARY OUTCOMES:
The degree of chronic pain using Brief Pain Inventory | 6 month post injection
  Brief Pain Inventory short form (BPI-SF) questionnaire. It is a nine item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, normal work, relations with other persons, sleep, and enjoyment of life on a 10 Point Scale
  BPI-SF was measured before, immediately after injection, 3 and 6 month post injection
The incidence of complication | 2 hours post-intervention
  complications as hypotension, headache and neck pain

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available upon a reasonable request from the corresponding author
Access Criteria: after the end of study for one year